CLINICAL TRIAL: NCT06957431
Title: A Phase I Trial of Zanzalintinib Combined With Eribulin in Advanced Liposarcoma and Leiomyosarcoma
Brief Title: Zanzalintinib Combined With Eribulin in Advanced Liposarcoma and Leiomyosarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202506154
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Advanced Leiomyosarcoma; Adipocytic Sarcoma; Advanced Liposarcoma
Keywords: Sarcoma; Eribulin; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Sarcoma | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 1 (starting dose): Zanzalintinib + Eribulin (Experimental): Patients will receive zanzalintinib 40 mg by mouth once daily on Days 1 through 21 and eribulin intravenously on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Zanzalintinib; Drug: Eribulin
- Dose Level 2: Zanzalintinib + Eribulin (Experimental): Patients will receive zanzalintinib 60 mg by mouth once daily on Days 1 through 21 and eribulin intravenously on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Zanzalintinib; Drug: Eribulin
- Dose Level -1: Zanzalintinib + Eribulin (Experimental): Patients will receive zanzalintinib 20 mg by mouth once daily on Days 1 through 21 and eribulin intravenously on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Zanzalintinib; Drug: Eribulin

INTERVENTIONS:
Drug: Zanzalintinib — Supplied by Exelixis, Inc.
  Other Names: XL092
Drug: Eribulin — 1.1 mg/m^2 dose.
  Other Names: Halaven

SUMMARY:
The investigators hypothesize that the combination of eribulin and zanzalintinib will be tolerable and lead to improved progression-free survival (PFS) as compared to eribulin alone based on historical data.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of unresectable or metastatic leiomyosarcoma or adipocytic sarcoma.
* Progressed on at least 1 line of prior therapy and have received no more than 4 lines of prior therapy.
* Measurable disease per RECIST 1.1.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Adequate bone marrow and organ function within 14 days before first dose of study treatment as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm without granulocyte colony-stimulating factor support within 2 weeks of collection
  * Platelets ≥ 100 K/cumm without transfusion within 2 weeks of collection
  * Hemoglobin ≥ 9.0 g/dL without transfusion within 2 weeks of collection
  * INR ≤ 1.5 x ULN and aPTT ≤ 1.2 x ULN; for subjects on Factor Xa inhibitors, this criterion does not apply.
  * Total bilirubin ≤ 1.5 x IULN (for subjects with Gilbert's disease, ≤ 3.0 x IULN)
  * AST(SGOT)/ALT(SGPT)/alkaline phosphatase (ALP) ≤ 3.0 x IULN (for subjects with documented bone metastasis, ALP ≤ 5.0 x IULN)
  * Serum albumin ≥ 2.8 g/dL
  * Serum creatine ≤ 1.5 x IULN or calculated creatinine clearance ≥ 40 mL/min by Cockcroft-Gault
  * UPCR ≤ 1 mg/mg (≤ 113.2 mg/mmol) creatinine
* Recovery to baseline or ≤ grade 1 from AEs, including immune-related AEs related to any prior treatments, unless AEs are clinically nonsignificant and/or stable on supportive therapy (e.g., physiological replacement of corticosteroid). Low-grade or controlled toxicities such as alopecia, ≤ grade 2 hypomagnesemia, ≤ grade 2 neuropathy are permitted.
* The effects of zanzalintinib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 186 days after last dose of zanzalintinib (for women) or 96 days after last dose of zanzalintinib (for men). Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Pure well-differentiated liposarcoma or low grade leiomyosarcoma.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Prior treatment with zanzalintinib.
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
* Radiation therapy for bone metastasis within 2 weeks before first dose of study treatment; any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Currently receiving any other investigational agents.
* Patients with untreated brain metastases. Patients with treated brain metastases are allowed if post-treatment brain-imaging after CNS-directed therapy shows no evidence of progression and disease is stable for at least 4 weeks before first dose of study treatment.

  * Note: eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of enrollment.
  * Note: base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to zanzalintinib or eribulin or other agents used in the study.
* Concomitant anticoagulation with warfarin or other vitamin-K antagonists, direct thrombin inhibitors, or antiplatelet agents (e.g. clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.
  * Note: subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer.
* Any complementary medications (e.g. herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study treatment.
* Uncontrolled, significant intercurrent or recent illness including, but not limited to:

  * Unstable or deteriorating cardiovascular disorders:

    * Congestive heart failure NYHA Class 3 or 4, or Class 2 or higher unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (e.g. ventricular flutter, ventricular fibrillation, Torsades de pointes).
    * Uncontrolled hypertension defined as sustained blood pressure > 140 mmHg systolic or > 90 mmHg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack), myocardial infarction, or other clinically significant arterial thrombotic and/or ischemic event within 6 months before first dose of study treatment.
    * Pulmonary embolism or deep vein thrombosis or prior clinically significant venous events within 3 months before first dose of study treatment.

      * Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.
      * Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the PI.
    * Prior history of myocarditis.
  * Gastrointestinal disorders, including those associated with a high risk of perforation or fistula formation:

    * Tumors invading the GI tract from external viscera
    * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis
    * Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months before first dose unless cause of obstruction is definitively managed and subject is asymptomatic.
    * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose.

      * Note: complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
    * Known gastric or esophageal varices.
    * Ascites, pleural effusion, or pericardial fluid requiring drainage in last 4 weeks.
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 mL) of red blood, or other history of significant bleeding (e.g. pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
* Symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed).
* Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta.

  * Note: subjects with intravascular tumor extension (e.g. tumor thrombus in renal vein on inferior vena cava) may be eligible following PI approval.
* Other clinically significant disorders that would preclude safe study participation.

  * Active infection requiring systemic treatment.

    * Note: prophylactic antimicrobial treatments (antibiotics, antimycotics, antivirals) are allowed.
  * Known infection with acute or chronic hepatitis B or C, known HIV or AIDS-related illness except for subjects meeting all of the following criteria:

    * On stable anti-retroviral therapy
    * CD4+ T cell count ≥ 200/μL
    * Undetectable viral load.

      * Note: HIV testing will be performed at screening if and as required by local regulation.
      * Note: to be eligible, participants taking strong or moderate CYP inhibitors (e.g. zidovudine, ritonavir, cobicistat, didanosine) or strong or moderate CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies must have been received for at least 4 weeks prior to the first dose.
      * Note: CD4+ T cell counts and viral load are monitored per standard of care by the local health provider.
  * Serious non-healing wound/ulcer/bone fracture.

    * Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
  * Malabsorption syndrome.
  * Pharmacologically uncompensated, symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ or allogeneic stem cell transplant.
* Major surgery (e.g. GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to first dose of study treatment. Prior laparoscopic surgeries (e.g. nephrectomy) within 4 weeks prior to first dose of study treatment. Minor surgery (e.g. simple excision, tooth extraction) within 5 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study treatment.

  * Note: fresh tumor biopsies should be performed at least 5 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 14 days per ECG before first dose of study treatment.

  * Note: triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
* History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Inability to swallow tablets or ingest a suspension either orally or by a NG or PEG tube.
* Other conditions which, in the opinion of the Investigator, would compromise the safety of the patient or the patient's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2033-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events experienced by participants | From start of treatment through 30 days after completion of treatment (estimated to be 25 months)
  Graded using CTCAE version 5.0.
Maximum tolerated dose (MTD)/recommended phase II dose (RP2D) | Through cycle 1 of treatment (each cycle is 21 days)
  The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. Dose escalations will proceed until the MTD has been reached or, if the MTD is not reached, until 6 patients have been treated successfully at the highest dose level (which will then be termed the recommended phase II dose (RP2D)).

SECONDARY OUTCOMES:
Overall response rate (ORR) by RECIST 1.1 | Through completion of treatment (estimated to be 24 months)
  * ORR is defined as number of patients with complete response (CR) or partial response (PR).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free survival (PFS) | 6 months from start of treatment
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Median Overall survival (OS) | Through completion of follow-up (estimated to be 7 years)
  - OS is defined as the duration of time from start of treatment to time of death.
Kaplan-Meier Estimate of Overall survival (OS) | 24 months from start of treatment
  - OS is defined as the duration of time from start of treatment to time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Mia C Weiss, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu